CLINICAL TRIAL: NCT05062083
Title: PET Imaging of Cyclooxygenases in Multiple Sclerosis
Brief Title: PET Imaging of Cyclooxygenase in Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to futility
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000483; 000483-M
Record Dates: First submitted 2021-09-29; First posted 2021-09-30 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: PET Imaging; Multiple Sclerosis; Neuroinflammation; Neurological Symptoms; Cyclooxygenases
MeSH Terms: conditions — Multiple Sclerosis; Neuroinflammatory Diseases; Neurologic Manifestations | interventions — (11C)-MC1; 11C-PS13; Ketoprofen; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with multiple sclerosis (Experimental): Participants had two brain positron emission tomography (PET) scan visits. In one visit, participants had a baseline [11C]PS13 scan followed by a second [11C]PS13 scan after blockade with ketoprofen 75 mg orally. In another visit, participants had baseline [11C]MC1 scan followed by a second scan with [11C]MC1 after blockade by a dose of celecoxib 600 mg orally. Participants receive injection of up to 20 millicurie (mCi) of [11C]PS13 or [11C]MC1 during each scan.
  Interventions: Drug: 11C-MC1; Drug: 11C-PS13; Drug: Ketoprofen; Drug: Celecoxib

INTERVENTIONS:
Drug: 11C-MC1 — Up to 20 mCi injected IV followed by PET scanning
Drug: 11C-PS13 — Up to 20 mCi injected IV followed by PET Scanning
Drug: Ketoprofen — Ketoprofen 75 mg orally once
Drug: Celecoxib — celecoxib 600 mg orally once

SUMMARY:
Background:

Multiple sclerosis (MS) is an autoimmune disease that has no cure. MRI is the main tool used in the study and treatment of people with MS. Tracers have been developed for cyclooxygenase-1 (COX-1) and cyclooxygenase-2 (COX-2), key enzymes that involved in neuroinflammation. Researchers want to explore the role inflammation plays in MS and see if COX-1 and COX-2 are measurable in the brains of people with the disease.

Objective:

To see if COX-1 and COX-2 are detectable in the brains of individuals with MS.

Eligibility:

People ages 18 and older with MS who are otherwise healthy.

Design:

Participants will be screened with their medical history and a physical exam. They will have an EKG to check the electrical activity of the heart.

Participants study involvement requires 3 to 5 visits and will last between 2 weeks and 4 months.

Participants will have two positron emission tomography (PET) scans of the brain for each tracer. Scans of the same tracer might occur on the same day or on separate days. A small amount of a radioactive chemical will be injected through an intravenous catheter. A needle will be used to guide a thin plastic tube into an arm vein. The needle will be removed. Only the catheter will be left in the vein. The PET scanner is shaped like a doughnut. Participants will lie on a bed that slides in and out of the scanner. They will wear a plastic mask molded to fit the head. The scan will last about 90 minutes for each tracer. Participants will receive the medication ketoprofen or celecoxib orally about 2 hours before the second scan.

Participants will have blood tests.

Participants must avoid certain medications a month prior to the PET scans.

DETAILED DESCRIPTION:
Study Description: This study will examine whether cyclooxygenase 1 (COX-1) and cyclooxygenase 2 (COX-2) are elevated in the brain of individuals with Multiple Sclerosis (MS)

Objectives: To determine whether COX-1 and COX-2 are detectable in the brains of individuals with MS.

Endpoints:

Primary endpoint: Calculation of COX-1 and COX-2 densities from [11C]PS13 and [11C]MC1 PET scans, respectively, using baseline scans and scans after blockade with ketoprofen and celecoxib, respectively.

Secondary endpoint: 1) Comparison of [11C]PS13 and [11C]MC1 specific uptake in different types of MS lesions (active, chronic active, inactive) and in normal white matter. 2) Comparison of [11C]PS13 and [11C]MC1 specific uptake in the brain lesions of the same subjects

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 years and older.
* Female participants of childbearing potential must be using a medically acceptable means of contraception.
* Able to provide informed consent.
* In good general health as evidenced by medical history and physical examination.
* Enrolled under University of Maryland in Baltimore (UMB) protocol HP-00079860 (In vivo assessment of meningeal inflammation and its clinical impact in multiple sclerosis by 7 Tesla MRI), P.I. Daniel Harrison and have agreed to contact for future research.

EXCLUSION CRITERIA:

* Any medical contraindication to the procedures performed in the study, or any current severe medical or psychiatric illness other than MS. This includes contraindications to Celecoxib, such as aspirin sensitive asthma, and contraindications to ketoprofen, such as hypersensitivity to ketoprofen or history of upper or lower gastrointestinal bleeding.
* Behavioral symptoms that would preclude the gathering of data for the study, or advanced disease such that subjects cannot provide assent.
* Clinically significant abnormalities on EKG or safety labs. This includes complete blood count (CBC); acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen); hepatic panel [alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin total, and bilirubin direct]; mineral panel (albumin, calcium, magnesium, phosphorus).
* MRI performed >180 days before or after the PET scan
* Have taken NSAIDs for two weeks prior to the PET scan. Have taken aspirin, corticosteroids (except for topical creams), or immunosuppressants (except for FDA approved disease-modifying therapy for MS) in the prior month.
* Have other major neurological or medical diseases that may cause cognitive dysfunction, such as structural brain diseases, metabolic diseases, paraneoplastic syndromes, infectious diseases, or other significant neurological abnormalities.
* Have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the patient and/or caregiver during the screening visit.
* Pregnancy
* HIV infection
* Be National Institute of Mental Health (NIMH) staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

Exclusion of Children

Because this protocol has more than minimal risk from radiation exposure without possibility of direct benefit, inclusion of children is not appropriate.

Exclusion of Pregnant or Breastfeeding Women

Pregnant women will be excluded because this protocol involves exposure to ionizing radiation. Lactating women will be excluded because radioisotopes may be excreted in milk.

Exclusion of Participants who are HIV Positive

Persons with HIV infection are excluded because HIV infection itself may cause neuroinflammation, and we wish to specifically study the effect of MS on neuroinflammation.

Exclusion of Participation of NIH Staff or family members of study team members NIH staff and family members of study team members may not be enrolled in this study.

INCLUSION OF VULNERABLE PARTICIPANT

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.This study will also comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule.
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol
Access Criteria: Biomedical Translational Research Information System (BTRIS)

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000483-M.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the seven participants who were consented to the study, two participants were screen failure.
Period: Overall Study
Arm/Group | Participants With Multiple Sclerosis
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Standard Uptake Value Ratio (SUVR) of Lesions With Injection of [11C]PS13
Description: Standard uptake value (SUV) was measured by averaging the SUV of all lesion voxels or tissue contralateral to lesion voxels in the PET image with injection of [11C]PS13. The SUVR was calculated by averaging the SUV ratio between lesion or tissue contralateral to lesion voxels and the caudate from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR)
  Brain lesions | 1.380 (0.112)
  Contralateral normal appearing brain tissues | 1.408 (0.109)

2. Primary Outcome: Standard Uptake Value Ratio (SUVR) of Lesions With Injection of [11C]MC1
Description: Standard uptake value (SUV) was measured by averaging the SUV of all lesion voxels or tissue contralateral to lesion voxels in the PET image with injection of [11C]MC1. The SUVR was calculated by averaging the SUV ratio between lesion or tissue contralateral to lesion voxels and the cerebellum from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR)
  Brain lesions | 1.455 (0.142)
  Contralateral normal appearing brain tissues | 1.594 (0.120)

3. Primary Outcome: Standard Uptake Value Ratio (SUVR) of Lesions With Injection of [11C]PS13 After Blockade With Ketoprofen
Description: Calculation of standard uptake value (SUV) by averaging the SUV of all lesion voxels or tissue contralateral to lesion voxels in the PET image with injection of [11C]PS13 after blockade with ketoprofen. Calculation of SUVR by averaging the SUV ratio between lesion or tissue contralateral to lesion voxels and the caudate from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR) | NA (NA) — Insufficient imaging signal above the lower limit of quantitation (LLOQ)

4. Secondary Outcome: Standard Uptake Value Ratio (SUVR) of Chronic Active Lesions With Injection of [11C]PS13
Description: Chronic active lesion is defined as the white matter lesion with paramagnetic outer rim in quantitative susceptibility maps (QSM). Standard uptake value (SUV) was measured by averaging the SUV of chronic active lesion voxels or contralateral normal appearing brain tissues in the [11C]PS13 PET image. The SUVR was calculated by averaging the SUV ratio between chronic active lesion or tissue contralateral to lesion voxels and the caudate from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR)
  Chronic active lesion | 1.424 (0.033)
  Contralateral normal appearing brain tissues | 1.455 (0.196)

5. Secondary Outcome: Standard Uptake Value Ratio (SUVR) of Chronic Active Lesions With Injection of [11C]MC1
Description: Chronic active lesion is defined as the white matter lesion with paramagnetic outer rim in quantitative susceptibility maps (QSM). Standard uptake value (SUV) was measured by averaging the SUV of chronic active lesion voxels or contralateral normal appearing brain tissues in the [11C]MC1 PET image. The SUVR was calculated by averaging the SUV ratio between chronic active lesion or tissue contralateral to lesion voxels and the cerebellum from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR)
  Chronic active lesion | 1.562 (0.080)
  Contralateral normal appearing brain tissues | 1.724 (0.143)

6. Primary Outcome: Standard Uptake Value Ratio (SUVR) of Lesions With Injection of [11C]MC1 After Blockade With Celecoxib
Description: Calculation of standard uptake value (SUV) by averaging the SUV of all lesion voxels or tissue contralateral to lesion voxels in the PET image with injection of [11C]MC1 after blockade with celecoxib. Calculation of SUVR by averaging the SUV ratio between lesion or tissue contralateral to lesion voxels and the cerebellum from 60-90 minutes after the start of the PET scan.
Time Frame: 60-90 minutes after the start of PET scan
Population: The analyses included only subjects who completed the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Participants With Multiple Sclerosis
Number analyzed (Participants) | 5
SUV Ratio (SUVR) | NA (NA) — Insufficient imaging signal above the lower limit of quantitation (LLOQ)

ADVERSE EVENTS:
Time Frame: Up to three days after each PET scan
Arm/Group | Participants With Multiple Sclerosis
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT05062083/Prot_SAP_000.pdf